CLINICAL TRIAL: NCT01116011
Title: A Phase I, Single-Centre, Randomised, Double-Blind, Placebo-controlled, Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD7268 When Given in Multiple Ascending Oral Doses in Japanese Healthy Male Subjects
Brief Title: Multiple Ascending Dose Study for AZD 7268 in Japanese Healthy Male Volunteers
Acronym: JMAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, AstraZeneca
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: D1151C00004
Record Dates: First submitted 2010-04-13; First posted 2010-05-04 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: Phase I; Japanese Healthy volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD7268 (Experimental)
  Interventions: Drug: AZD7268
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7268 — Capsule, Oral, BID
  Arms: AZD7268
Drug: Placebo — Capsule, Oral, BID
  Arms: Placebo

SUMMARY:
This is a multiple ascending dose study (MAD) in the Japanese population with AZD7268. This MAD study will evaluate the safety, tolerability and pharmacokinetics of orally administered AZD7268 after multiple ascending doses.

ELIGIBILITY:
Inclusion Criteria:

* Provision of Informed Consent
* Healthy male subjects, with suitable veins for cannulation or repeated venipuncture

Exclusion Criteria:

* Inability to understand or cooperate with given information
* Any positive result on screening for human immune deficiency virus (HIV), Hepatitis B, Hepatitis C and syphilis test
* History of seizure (including infant febrile seizures) or family history of seizure

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Investigate the safety and tolerability of AZD7268 by Adverse Events. | From first dosing throughout the treatment period and including the follow-up period

SECONDARY OUTCOMES:
Characterize the PK parameters(Cmax, AUC,t1/2) of AZD7268 by assessment of drug concentrations in plasma | Blood samples will be taken from pre-dose until 48 hours post last dose
Characterize the PK parameters (CLr, Ae) of AZD7268 by assessment of drug concentrations in urine | Urine samples will be taken from post first dose until 48 hours post last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Tomoe Fujita, Principal Investigator — Kitasato University East Hospital, Kanagawa, Japan
Locations (1):
- Research Site, Kanagawa, Sagamihara, Japan